CLINICAL TRIAL: NCT04129151
Title: Phase 2 Trial of Palbociclib and Ganitumab in Patients With Relapsed or Refractory Ewing Sarcoma
Brief Title: Palbociclib + Ganitumab In Ewing Sarcoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study closed early due to discontinuation of ganitumab supply.
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: 1 Million 4 Anna Foundation (Other); Carson Sarcoma Foundation (Other); Teaming up to Fight Childhood Cancer (Other); ChemoWarrior: the eli sidler foundation (Unknown); i-ROK Foundation (Other); Rutledge Cancer Foundation (Other); Alan B. Slifka Foundation (Other)
Responsible Party: Principal Investigator, David S Shulman, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-373
Record Dates: First submitted 2019-10-14; First posted 2019-10-16 (Actual); Results first posted 2024-07-17 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Ewing Sarcoma; Ewing's Sarcoma Recurrent
Keywords: Relapsed or refractory Ewing sarcoma; Solid Tumor, Childhood; Sarcoma; Ewing sarcoma
MeSH Terms: conditions — Sarcoma, Ewing; Recurrence; Sarcoma | interventions — palbociclib; ganitumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- PALBOCICLIB and GANITUMAB (Experimental): Participants receive up to 12 cycles of therapy (cycle duration=28 days).
  * Palbociclib: Oral, 100mg, daily on days 1-21
  * Ganitumab: Intravenous, 18mg/kg, days 1, 15
  Per protocol, participants were monitored for dose-limiting toxicity over cycle one according to an interim safety analysis. The safety monitoring rule was triggered after 3 patients had enrolled, prompting an amendment according to Contingency Plan A which was a reduction of the palbociclib dose from 125mg (days 1-21).
  Interventions: Drug: Palbociclib; Drug: Ganitumab

INTERVENTIONS:
Drug: Palbociclib — Oral, per protocol pre determined dosage, once a day for 21 days
  Other Names: Ibrance®
Drug: Ganitumab — -Intravenous, per protocol predetermined dosage, twice per cycle
  Other Names: AMG-479

SUMMARY:
This research study is designed to study the combination of two drugs, palbociclib and ganitumab, as a potential treatment for Ewing sarcoma.

The names of the study drugs involved in this study are:

* Palbociclib
* Ganitumab

DETAILED DESCRIPTION:
This research study involves participants taking a medicine that inhibits proteins in cancer cells called CDK4 and CDK6 (palbociclib) in combination with a medicine that inhibits a protein called IGF-1R (ganitumab). This study is designed to see if these drugs are safe when given together and whether they are effective in treating Ewing sarcoma.

This research study is a Phase II clinical trial. Phase II clinical trials test the safety and effectiveness of an investigational drug or drug combination to learn whether the drug(s) works in treating a specific disease. "Investigational" means that the drug or combination is being studied.

The U.S. Food and Drug Administration (FDA) has not approved ganitumab as a treatment for any disease.

The U.S. Food and Drug Administration (FDA) has not approved palbociclib for this specific disease but it has been approved for another cancer.

This research study is:

* Testing whether palbociclib and ganitumab are safe when given together and effective in treating Ewing sarcoma.
* Testing markers in the blood and in tumor tissue to see if there are certain features of the tumor that may indicate this combination of drugs is effective or not effective

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 12 years and ≤ 50 years at time of enrollment.
* Karnofsky performance status ≥ 50% for patients ≥16 years of age and Lansky ≥ 50% for patients <16 years of age (see Appendix A)
* Disease Requirement: Participants must have relapsed or refractory Ewing sarcoma with:

  * RECIST measurable disease at study entry, including at least one RECIST measurable site that has either not been previously radiated or that has had progression after prior radiotherapy;
  * Histologic diagnosis consistent with Ewing sarcoma or PNET; and
  * Molecular evidence of translocation involving EWSR1 or FUS (also known as TLS), such as FISH, RT-PCR, or next generation sequencing. If the translocation partner is known it must be of the ETS family (i.e. FLI1 or ERG).
* Participants must have disease for which standard curative or palliative measures do not exist or are no longer effective.
* Patients must have fully recovered (Common Terminology Criteria for Adverse Events [CTCAE] version 5 Grade ≤1) from the acute toxic effects of all prior anti-cancer therapy except organ function as noted in Section 3.1.6. Patients must meet the following minimum washout periods prior to enrollment:
* Myelosuppressive chemotherapy: At least 14 days after the last dose of myelosuppressive chemotherapy (42 days for nitrosourea or mitomycin C).
* Radiotherapy:

  * At least 14 days after local palliative XRT (small port);
  * At least 90 days must have elapsed after craniospinal XRT or if >50% radiation of pelvis;
  * At least 6-months must have elapsed following TBI or thoracic radiation involving the lungs;
  * At least 42 days must have elapsed if other substantial bone marrow radiation;
* Small molecule biologic therapy: At least 7 days following the last dose of a biologic agent. For agents with known adverse events occurring beyond 7 days, this duration must be extended beyond the time in which adverse events are known to occur. If extended duration is required, this should be discussed and approved by the study chair.
* Monoclonal antibody: At least 21 days must have elapsed after the last dose of antibody.
* Myeloid growth factors: At least 14 days following the last dose of long-acting growth factor (e.g. Neulasta®) or 7 days following short-acting growth factor.
* Immunotherapy: At least 4 weeks since the completion of immunotherapy (e.g. tumor vaccines) aside from monoclonal antibodies with immune effects covered under Section 3.1.5.4.
* Stem Cell Infusion or Cellular Therapies: The patient must have no evidence of graft versus host disease and at least 42 days must have elapsed after transplant, stem cell infusion, or cellular therapy.
* Major Surgery: At least 2 weeks from prior major surgical procedure. Note: Biopsy and central line placement/removal are not considered major surgery.
* CDK4/6 and IGF-1R inhibitors: The participant must not have received a prior CDK4/6 inhibitor. Prior therapy with IGF-1R inhibitor is allowed if the patient did not relapse while on IGF-1R therapy. Patients must not have received prior therapy with a combination of CDK4/6 inhibitor and IGF-1R inhibitor.
* Participants must have normal organ function as defined below.
* Hematologic Requirements for Subjects without Known Bone Marrow Involvement by Disease:

  * Absolute neutrophil count ≥ 1000 /uL
  * Hemoglobin ≥ 8 g/dL (transfusion allowed)
  * Platelets ≥100,000 /uL and transfusion independent, defined as not receiving a platelet transfusion for at least 7 days prior to CBC documenting eligibility.
* Hematologic Requirements for Subjects with Bone Marrow Involvement by Disease as Demonstrated on Clinically-Indicated Bone Marrow Biopsy:

  * Absolute neutrophil count >750 /uL
  * Hemoglobin ≥ 8 g/dL (transfusion allowed)
  * Platelets ≥50,000 /uL and transfusion independent, defined as not receiving a platelet transfusion for at least 7 days prior to CBC documenting eligibility.
  * Not known to be refractory to platelet or red cell transfusions.
* Hepatic Function:

  * Total bilirubin ≤ 1.5 x upper limit of normal for age Patients with Gilbert's syndrome with a total bilirubin < 2 x upper limit of normal for age and a direct bilirubin within normal limits are permitted.
  * ALT (SGPT) ≤ 135 U/L For the purpose of this study, the ULN for ALT is 45 U/L
  * AST (SGOT)≤ 90 U/L For the purpose of this study, the ULN for AST is 90 U/L
  * Serum albumin ≥ 2 g/dL
* Renal Function:

  -- A serum creatinine based on age/gender as follows: Maximum Serum Creatinine (mg/dL) Male Female
  * 12 to < 13 years 1.2 1.2
  * 13 to < 16 years 1.5 1.4
  * ≥ 16 years 1.7 1.4 Or
* Creatinine clearance ≥ 70 mL/min/1.73 m2 for participants with creatinine levels above institutional normal.
* Adequate Cardiac Function: QTc ≤ 480 msec on ECG
* Adequate GI Function: Diarrhea < grade 2 by CTCAE version 5
* Adequate Metabolic Function: Fasting glucose ≤ 160 mg/dL (or < 8.9 mmol/L) without the use of antihyperglycemic agents. If random glucose ≤ 160 mg/dL (or ≤ 8.9 mmol/L), fasting value does not need to be obtained.
* Additional Agent-Specific Requirements

  * Patients must be able to swallow capsules.
  * For patients with CNS metastatic disease, any baseline neurologic deficits (including seizure) must be stable for at least one week prior to study enrollment.
* Ability to understand and/or the willingness of the patient (or parent or legally authorized representative, if minor) to provide informed consent, using an institutionally approved informed consent procedure.

Exclusion Criteria:

* Patients must not be receiving any of the following concomitant medications:

  -- Pharmacologic doses of systemic corticosteroids unless for CNS metastatic disease. For patients with CNS metastatic disease receiving corticosteroids, they should be on a stable or decreasing dose over the 7 days prior to registration Section 3.1.6.7 of protocol document. For all patients, receipt of systemic physiologic replacement steroids, topical and/or inhaled corticosteroids is acceptable.
* Patients receiving medications that are strong inhibitors or inducers of CYP3A4 within 7 days of enrollment (refer to Appendix B, Table 10 for prohibited medications)
* Patients receiving medications that cause significant QTc prolongation as outlined in Table 12 of Appendix B.
* Patients who have had tumor molecular testing with sequencing of the RB1 gene and were found to have RB1 mutation or loss will be excluded.
* Patients with a history of pneumonitis will be excluded.
* Pregnant participants will not be entered on this study given that the effects of palbociclib and ganitumab on the developing human fetus are unknown.
* Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with palbociclib and ganitumab, breastfeeding mothers are not eligible.
* Participants of child-bearing or child-fathering potential must agree to use adequate contraception (hormonal birth control; intrauterine device; double barrier method; or total abstinence) throughout their participation, including up until 30 days after last dose of palbociclib or ganitumab, whichever was administered last.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to palbociclib or ganitumab.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Participants with a personal history of any of the following: syncope due to an intrinsic cardiac etiology (note that syncope due to vasovagal episodes or dehydration/orthostasis would NOT exclude a participant), pathologic ventricular arrhythmias (including, but not limited to, ventricular tachycardia and ventricular fibrillation), or sudden cardiac arrest.
* Patients with known HIV, hepatitis B, and/or hepatitis C (testing not required as part of screening).
* Patients with a known history of type 1 or type 2 diabetes mellitus.
* Patients with gastrointestinal disease or disorder that could interfere with absorption of palbociclib, such as bowel obstruction or inflammatory bowel disease.
* Patients < 40 kg will be excluded given use of palbociclib at non-weight / non-BSA based flat dosing.

Ages: 12 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2019-12-05 (Actual); Primary Completion 2022-12-15 (Actual); Study Completion 2022-12-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Shulman, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (3):
- United States (3):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Boston Children's Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: contact Sponsor Investigator or designee. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu

REFERENCES:
- [Result] Shulman DS, Merriam P, Choy E, Guenther LM, Cavanaugh KL, Kao PC, Posner A, Bhushan K, Fairchild G, Barker E, Klega K, Stegmaier K, Crompton BD, London WB, DuBois SG. Phase 2 trial of palbociclib and ganitumab in patients with relapsed Ewing sarcoma. Cancer Med. 2023 Jul;12(14):15207-15216. doi: 10.1002/cam4.6208. Epub 2023 Jun 12. PMID 37306107

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were enrolled between December 2019 and August 2021.
Groups:
- PALBOCICLIB and GANITUMAB: This is a single arm, open-label, phase 2 study of ganitumab and palbociclib. Patients started treatment with standard dosing (Palbociclib 125 mg on days 1-21 and ganitumab 18 mg/kg on days 1 and 15 of a 28-day cycle). Safety stopping rules were used to monitor for toxicity of this novel combination therapy. Participants received up to 12 cycles of therapy in a single cohort.
  The first 3 participants started treatment at standard dosing (Palbociclib 125 mg on days 1-21 and ganitumab 18 mg/kg on days 1 and 15 of a 28-day cycle). After 2 initial patients experienced dose limiting toxicity, safety stopping rules were triggered and the starting palbociclib dose was reduced to 100 mg on days 1-21 (ganitumab dose was not changed). The subsequent 7 participants were treated at the reduced starting dose (Palbociclib 100 mg on days 1-21 and ganitumab 18 mg/kg on days 1 and 15 of a 28-day cycle). This study did not include formal dose escalation given both agents had previously established recommended phase 2 dosing.
Period: Overall Study
Arm/Group | PALBOCICLIB and GANITUMAB
Started | 10
Completed | 1
Not Completed | 9
Not completed — Adverse Event | 1
Not completed — Disease Progression | 7
Not completed — Study closure | 1

BASELINE CHARACTERISTICS:
Groups:
- PALBOCICLIB and GANITUMAB: Participants receive up to 12 cycles of therapy (cycle duration=28 days).
  Palbociclib: Oral, 100mg, daily on days 1-21 Ganitumab: Intravenous, 18mg/kg, days 1, 15
  Per protocol, participants were monitored for dose-limiting toxicity over cycle one according to an interim safety analysis. The safety monitoring rule was triggered after 3 patients had enrolled, prompting an amendment according to Contingency Plan A which was a reduction of the palbociclib dose from 125mg (days 1-21).
Arm/Group | PALBOCICLIB and GANITUMAB
Number analyzed (Participants) | 10
Age, Continuous [Median (Full Range); unit: Years] | 25.7 [12.3 to 40.1]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 7
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 8
  More than one race | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Non-Hispanic | 10
  Hispanic | 0
Primary site at diagnosis [Count of Participants; unit: Participants]
  Bone | 8
  Soft tissue | 2
Primary site at diagnosis [Count of Participants; unit: Participants]
  Femur | 3
  Iliac | 2
  Gluteal soft tissue | 2
  Scapula | 1
  Tibia | 1
  Thoracic vertebra | 1
Translocation [Count of Participants; unit: Participants]
  EWSR1/FLI1 | 5
  EWSR1-translocation by FISH | 5
Prior IGF - 1R therapy [Count of Participants; unit: Participants]
  No | 10
  Yes | 0
Stage at diagnosis [Count of Participants; unit: Participants]
  Localized | 4
  Metastatic | 6

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: ORR was defined as the percentage of participants achieving complete response (CR) or partial response (PR) on treatment based on RECIST 1.1 criteria. Per RECIST 1.1 for target lesions: CR is complete disappearance of all target lesions and PR is at least a 30% decrease in the sum of longest diameter (LD) of target lesions, taking as reference baseline sum LD. PR or better overall response assumes at a minimum incomplete response/stable disease (SD) for the evaluation of non-target lesions and absence of new lesions.
Time Frame: Participants were followed up to 10.8 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | PALBOCICLIB and GANITUMAB
Number analyzed (Participants) | 10
percentage of participants | 0 [0 to 30]

2. Primary Outcome: Grade 3/4 Treatment-Related Toxicity Rate
Description: The proportion of participants who experienced a maximum grade 3 or 4 treatment-related adverse event based on the Common Toxicity Criteria for Adverse events Version 5.0 (CTCAEv5) as reported on case report forms
Time Frame: Participants were followed up to 11.8 months.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | PALBOCICLIB and GANITUMAB
Number analyzed (Participants) | 10
proportion of participants | 0.8 [0.44 to 0.97]

3. Secondary Outcome: 6-month Progression Free Survival (PFS6)
Description: PFS6 is the percent probability estimate at 6 months based on the Kaplan-Meier method. PFS is defined as the duration of time from study entry to documented disease progression (PD) requiring removal from the study or death. Participants alive without PD were censored at the earliest of the date of the last disease evaluation or start of new anticancer therapy. Per RECIST 1.1 for target lesions: PD is at least a 20% increase in sum LD, taking as reference the smallest sum on study with at least 5 mm absolute increase. For non-target lesions, progression-free means no new lesions or unequivocal progression on existing non-target lesions or not evaluated.
Time Frame: Participants were followed up to 6 months.
Measure: Number (95% Confidence Interval); unit: Percent Probability
Arm/Group | PALBOCICLIB and GANITUMAB
Number analyzed (Participants) | 10
Percent Probability | 30 [1.6 to 58.4]

4. Secondary Outcome: 6-month Overall Survival (OS6)
Description: OS6 is the percent probability estimate at 6 months based on the Kaplan-Meier method. Overall survival was defined as the time from study enrollment to death. Participants alive were censored at the last date of contact (including lost-to-follow-up) or at the date of withdrawal of consent, if relevant.
Time Frame: Participants were followed up to 6 months.
Measure: Number (95% Confidence Interval); unit: Percent Probability
Arm/Group | PALBOCICLIB and GANITUMAB
Number analyzed (Participants) | 10
Percent Probability | 80 [55.1 to 100]

ADVERSE EVENTS:
Time Frame: Participants were followed for AEs up to 11.8 months and survival up to 2 years.
Description: Serious adverse events were defined per protocol section (7.6). All remaining adverse events were classified as other adverse events. Maximum grade per toxicity type is presented.
Arm/Group | PALBOCICLIB and GANITUMAB
All-Cause Mortality (participants affected / at risk) | 6/10
Serious Adverse Events (participants affected / at risk) | 1/10
Other Adverse Events (participants affected / at risk) | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PALBOCICLIB and GANITUMAB (N=10)
Non-Cardiac Chest Patin (General disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PALBOCICLIB and GANITUMAB (N=10)
Anemia (Blood and lymphatic system disorders) | 8
Eosinophilia (Blood and lymphatic system disorders) | 1
Sinus bradycardia (Cardiac disorders) | 1
Sinus tachycardia (Cardiac disorders) | 4
Hypothyroidism (Endocrine disorders) | 1
Vision decreased (Eye disorders) | 1
Abdominal distension (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 3
Constipation (Gastrointestinal disorders) | 3
Diarrhea (Gastrointestinal disorders) | 7
Dyspepsia (Gastrointestinal disorders) | 1
Flatulence (Gastrointestinal disorders) | 2
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1
Mucositis oral (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 4
Oral pain (Gastrointestinal disorders) | 1
Toothache (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 3
Edema limbs (General disorders) | 1
Fatigue (General disorders) | 7
Fever (General disorders) | 2
Gait disturbance (General disorders) | 1
General disorders and administration site conditions - Other, specify (General disorders) | 1
Non-cardiac chest pain (General disorders) | 4
Pain (General disorders) | 4
Immune system disorders - Other, specify (Immune system disorders) | 2
Gum infection (Infections and infestations) | 1
Infections and infestations - Other, specify (Infections and infestations) | 1
Bruising (Injury, poisoning and procedural complications) | 2
Infusion related reaction (Injury, poisoning and procedural complications) | 1
Wound complication (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 2
Alkaline phosphatase increased (Investigations) | 2
Aspartate aminotransferase increased (Investigations) | 2
Blood bicarbonate decreased (Investigations) | 2
Creatinine increased (Investigations) | 4
Hemoglobin increased (Investigations) | 1
Investigations - Other, specify (Investigations) | 1
Lymphocyte count decreased (Investigations) | 4
Neutrophil count decreased (Investigations) | 9
Platelet count decreased (Investigations) | 9
Weight loss (Investigations) | 1
White blood cell decreased (Investigations) | 10
Anorexia (Metabolism and nutrition disorders) | 5
Hyperglycemia (Metabolism and nutrition disorders) | 3
Hyperkalemia (Metabolism and nutrition disorders) | 4
Hypermagnesemia (Metabolism and nutrition disorders) | 3
Hyperphosphatemia (Metabolism and nutrition disorders) | 4
Hypocalcemia (Metabolism and nutrition disorders) | 2
Hypomagnesemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 2
Hypophosphatemia (Metabolism and nutrition disorders) | 4
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 4
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1
Muscle cramp (Musculoskeletal and connective tissue disorders) | 1
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Concentration impairment (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 1
Headache (Nervous system disorders) | 5
Muscle weakness right-sided (Nervous system disorders) | 1
Peripheral motor neuropathy (Nervous system disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 2
Syncope (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 2
Depression (Psychiatric disorders) | 4
Insomnia (Psychiatric disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 2
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 1
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 2
Urticaria (Skin and subcutaneous tissue disorders) | 1
Hot flashes (Vascular disorders) | 1
Hypertension (Vascular disorders) | 2
Hypotension (Vascular disorders) | 3

LIMITATIONS AND CAVEATS:
The study terminated before full accrual.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-05-10): https://cdn.clinicaltrials.gov/large-docs/51/NCT04129151/Prot_SAP_001.pdf